CLINICAL TRIAL: NCT06556966
Title: A Phase Ⅰ, Randomized, Double-blind, Placebo-controlled, Single Dose Ascending Study to Assess the Safety, Tolerability, and Pharmacokinetics of LPM787000048 Maleate Sustained-release Tablet (LY03020) in Chinese Healthy Adult Subjects
Brief Title: A Study Assessing the Safety and Tolerability of LY03020 in Chinese Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LY03020/CT-CHN-101
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia; Alzheimer's Disease Psychosis
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LY03020 (Experimental): Subjects will take single-dose LY03020 on Day 1
  Interventions: Drug: LY03020
- Placebo (Sham Comparator): Subjects will take single-dose Placebo on Day 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY03020 — LY03020 for one single dose
  Other Names: LPM787000048 Maleate sustained-release tablet
  Arms: LY03020
Drug: Placebo — Placebo for one single dose
  Other Names: Placebo of LPM787000048 Maleate sustained-release tablet
  Arms: Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, ascending single oral dose study to assess the safety, tolerability, and pharmacokinetics of LY03020 in Chinese healthy adult subjects.

DETAILED DESCRIPTION:
The study will set 2.5mg, 5mg, 10mg, 20mg, 40mg, 60mg, 80mg and 100mg, a total of 8 dose groups. Qualified subjects were enrolled in site at D-1 ( 1 day before administration ) and randomized.The subjects should fast for at least 10 hours before medication administration, with no restrictions on water intake. The subjects will be required to orally take LY03020 or a placebo on an empty stomach upon waking on D1 (the day of medication administration). From D1 to D7, they will undergo safety assessments and PK biological sample collection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects sign informed consent voluntarily.
* Male or female aged 18 to 45 years.
* Body weight ≥ 50.0 kg for male and ≥ 45.0 kg for female, and male or female greater than or equal to 18.5 but less than 26.0 kg/m2 of body mass index (BMI).

Exclusion Criteria:

* Subjects have any clinically significant medical condition or chronic disease.
* Subjects experienced a history of keratopathy, fundus disease, increased intraocular pressure,or angle-closure glaucoma.Subjects have a abnormal and clinically significant test for ophthalmic examination during screening.
* Subjects with condition that may interfere with the drug absorption, distribution, metabolism and excretion significantly.
* Subjects had a history of surgery within 3 months prior to administration, or had not recovered, or have a surgical plan during the study.
* Subjects have any clinically significant abnormal vital signs, laboratory values, and ECGs.
* Subjects have used any of nonprescription drugs within 7 days or prescription drugs within 28 days prior to administration.
* Subjects have a history of allergic diseases, or allergic to any substance contained in the formulation
* Subjects have a positive test for HBsAg, HCV-Ab, HIV-Ab, or syphilis serum reaction.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-02-13 (Actual); Study Completion 2025-02-13 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) | up to144 hours
  Percentage of adverse events

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) of LPM787000048 in plasma | up to144 hours
  Subject blood samples will be collected at 17 time points and pharmacokinetic parameters will be calculated.
Time to maximum observed concentration (Tmax) of LPM787000048 in plasma | up to144 hours
  Subject blood samples will be collected at 17 time points and pharmacokinetic parameters will be calculated.
Area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) of LPM787000048 in plasma | up to144 hours
  Subject blood samples will be collected at 17 time points and pharmacokinetic parameters will be calculated.
Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUC0-t) of LPM787000048 in plasma | up to144 hours
  Subject blood samples will be collected at 17 time points and pharmacokinetic parameters will be calculated.
Apparent terminal elimination half-life (t1/2) of LPM787000048 in plasma | up to144 hours
  Subject blood samples will be collected at 17 time points and pharmacokinetic parameters will be calculated.
Apparent volume of distribution（Vz/F） of LPM787000048 in plasma | up to144 hours
  Subject blood samples will be collected at 17 time points and pharmacokinetic parameters will be calculated.
Apparent total body clearance (CL/F) of LPM787000048 from plasma | up to144 hours
  Subject blood samples will be collected at 17 time points and pharmacokinetic parameters will be calculated.

OTHER OUTCOMES:
Quantitatively determine the concentration of LPM787000048 and major metabolites (if applicable) in urine and calculate the cumulative excretion ratio in urine. | up to144 hours
  One dose group will be selected for metabolite identification.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Wang, Principal Investigator — Beijing AnDing Hospital Capital Medical University
Locations (1):
- Beijing AnDing Hospital Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No